CLINICAL TRIAL: NCT03206008
Title: The Effect of Intraoperative Magnesium Sulfate Infusion on the Postoperative Recovery After Outpatient Surgery
Brief Title: The Effect of Intraoperative Magnesium Sulfate Infusion on the Postoperative Recovery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: hard to get an informed concent because of small number of indiaiton of surgery
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, LEE YEA JI, clinical professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B-1608-360-006
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal saline group (Placebo Comparator): after loading normal saline 100cc in 10-20 minutes, continuous infusion of normal saline until the end of surgery
  Interventions: Drug: Normal saline
- Magnesium group (Active Comparator): after loading magnesium sulfate dosing 50 mg/kg (100cc) in 10-20 minutes, continuous infusion of magnesium sulfate 15 mg/kg/h until the end of surgery
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate
  Arms: Magnesium group
Drug: Normal saline — Placebo
  Arms: Normal saline group

SUMMARY:
Evaluating analgesic effect of intraoperative magnesium sulfate infusion in the outpatient surgery case

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-65 year-old-patient (ASA I-II) who are planned to undergoing day surgery

Exclusion Criteria:

* ASA class ≥ III
* suspected imbalance of electrolyte
* myocardial damage or conduction delay
* myasthenia gravis or other neuromuscular disease
* impaired renal function
* already using any type of analgesia
* denial of participating in the study or not giving the informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
severity of postoperative pain | 1 hour interval
  checking the postoperative pain in score at the recovery room and outpatient surgery center

CONTACTS AND LOCATIONS:
Overall Officials: SangHwan Do, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, department of Anesthesia and pain, Seongnam, Gyenggo-do, South Korea

IPD SHARING:
Plan to Share IPD: No